# Statistical Analysis Plan

PROTOCOL NUMBER: 1200-0322

PROTOCOL TITLE : J-REGISTER

<u>Japanese Real-world</u> data for treatment of afatinib ( $\underline{GI}$ otrif®) in first-line setting and  $\underline{S}$ ubsequent  $\underline{T}$ herapies for patients with advanced  $\underline{EGFR}$  mutation-positive lung adenocarcinoma

**AUTHOR:** 

VERSION NUMBER AND DATE: <V1.0; 07 DEC 2022>

Document: \jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text

Author: Version Number: 1.0

Version Date: 07 DEC 2022

Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to

. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan <V1.0, 07 DEC 2022)> for J-REGISTER<1200-0322>.

| | Name | Signature | Date |
|-----------|-------------------------|--------------------------|------|
| Author: | | この文書を承認す<br> 2022年12月7日 | |
| Position: | <b>Statistical Team</b> | (ST) | |
| Company: | | | |

Document: \\jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text

Author: Author: Version Date: 07 DEC 2021

Reference: RWI\_WI\_BIOS0015

Effective Date: 05Jan2018

Template No.: RWI\_TP\_BIOS0013 Revision 1

# **MODIFICATION HISTORY**

| Unique | Date of the | Author | Significant Changes from |
|------------|-------------|--------|--------------------------------|
| Identifier | Document | | Previous Authorized Version |
| for this | Version | | |
| Version | | | |
| 1.0 | 2022/12/07 | | Not Applicable – First version |

Document: \jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Effective Date: 15Jun2018

# TABLE OF CONTENTS

| | | OCOL TITLE :J-REGISTER | | |
|---|---|---|---|---|
| | Japan | ese REal-world data for treatment of a | | |
| | | and Subsequent Therapies for patien | ts with advanced EGF | R mutation- |
| | | positive lung adenocarcinoma | | 1 |
| 1. | ABB | REVIATIONS | ••••• | 6 |
| <b>2.</b> | INTE | RODUCTION | ••••• | 8 |
| <b>3.</b> | STUI | DY OBJECTIVES AND OUTCOMI | ES | 8 |
| | 3.1 | Primary Outcome | | 8 |
| | 3.2 | Secondary Outcomes | | 9 |
| | 3.3 | Safety Outcome | | 9 |
| 4. | STU | DY DESIGN | ••••• | 9 |
| | 4.1 | General Description | | 9 |
| | 4.2 | Schedule of Events | | 9 |
| | 4.3 | Changes to Analysis from Protocol. | | 10 |
| <b>5.</b> | PLA] | NNED ANALYSES | ••••• | 10 |
| | 5.1 | Interim Analysis | | 10 |
| | 5.2 | Final Analysis | | 11 |
| <b>6.</b> | ANA | LYSIS SETŠ | | |
| | 6.1 | All Subjects Enrolled [ENR] Set | | 11 |
| | 6.2 | Analysis Set | | |
| 7. | GEN | ERAL CONSIDERATIONS | ••••• | 12 |
| | 7.1 | Censoring rule | | 12 |
| | 7.2 | Software Version | | |
| 8. | STA | FISTICAL CONSIDERATIONS | ••••• | |
| | 8.1 | Statistical Tests and Confidence Inte | ervals | |
| | 8.2 | Missing data | | |
| | 8.3 | Examination of Subgroups | | |
| 9. | OUT | PUT PRESENTATIONS | ••••• | 14 |
| <b>10.</b> | DISP | OSITION AND WITHDRAWALS. | ••••• | 15 |
| 11. | DEM | OGRAPHIC AND OTHER BASEL | INE CHARACTERI | ISTICS15 |
| | 11.1 | Derivations | | 16 |
| Doc | ument: | \jptok-sfs02\data1\PROJ\Boehringer\NZA72 | 2277_Biostatistics\Document | ation\SAP\SAP_text |
| Autl | hor: | | Version Number: | 1.0 |
| Ten | nplate N | o.: RWI_TP_BIOS0013 Revision 1 | Re | eference: RWI_WI_BIOS0015 |

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

. and



# Statistical Analysis Plan

| <b>12.</b> | STUDY MEDICATION EXPOSURE | 16 |
|---|---|---|
| | 12.1 Derivations | 16 |
| 13. | IF AFATINIB THERAPY IS ONGOING AND 'STOP DATE' IS BLANK, THEN 'LAST CONFIRMATION DATE' IS USED AS 'STOP DATE'. | |
| | OUTCOMES | 17 |
| | 13.1 Primary outcome | 17 |
| | 13.2 Secondary outcomes | 17 |
| 14. | SAFETY OUTCOMES | |
| 15. | REFERENCES | 17 |

Document: \jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

#### 1. ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event

AESI Adverse Event of Special Interest
ATC Anatomical Therapeutic Chemical

BI Boehringer Ingelheim

CI Confidence Interval

CRO Contract Research Organisation

EC Ethics Committee

eCRF Electronic Case Report Form

EDC Electronic Data Capture

EGFR Epidermal Growth Factor Receptor

EGFR-TKI Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor

eTMF Electronic Trial Master File

HR Hazard Ratio

ICF Informed Consent Form

IRB Institutional Review Board

ISF Investigator Site File

LL3 LUX-Lung 3 study

NBI Nippon Boehringer Ingelheim

NIS Non-Interventional Study

NSCLC Non-Small Cell Lung Cancer

 $\label{locument: locument} Document: $$ \ \\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text $$$ 

\_\_\_\_\_

Version Number:


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Author:

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

1.0



OS Overall Survival

PD Progressive Disease

PFS Progression Free Survival

PS Performance Status

SAE Serious Adverse Event

SAP Statistical Analysis Plan

SOP Standard Operating Procedures

TMF Trial Master File

TOT Time on Treatment

TOT1 First-line TOT

TTF Time-to-Treatment Failure

TTP Time to Progression

UMIN University hospital Medical Information Network

Document: \jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

#### 2. INTRODUCTION

This statistical analysis plan (SAP) describes the rules and conventions to be used in the analysis and presentation. It describes the data to be summarized and analyzed, including specifications of the statistical analyses to be performed.

This SAP is based on protocol version 1.0, dated 2020/09/04 and case report forms (CRFs) ver.6.0, dated 2021/03/08.

All planned analyses identified in this SAP will be performed by Real-World Evidence Solutions (RWES) Biostatistics following Database Lock.

#### 3. STUDY OBJECTIVES AND OUTCOMES

The primary objective is to confirm Time on Treatment (TOT) related to afatinib treatment as the first-line therapy (TOT1) in patients with EGFR mutation-positive NSCLC. The observation in the real-world setting of the time from the start of the first-line afatinib until the end of subsequent treatment in this study will provide insights on the sequence of treatment for patients. The Japanese healthcare system will enable this study to evaluate multiple treatment options after afatinib treatment.

## 3.1 Primary Outcome

The primary outcome of this study is TOT with afatinib in TOT1. This will be assessed as the time from the start of afatinib (Giotrif®) as first-line treatment until the end of afatinib treatment or death date by any cause, which occurs first.

Document: \\jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text

Author: Version Number:


1.0

Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018



- TOT from the start of afatinib until end of subsequent therapies in the second-line setting or death by any cause, whichever occurs first
- TOT from start of the second-line treatment until end of the second-line treatment or death by any case (TOT2), whichever occurs first
- OS and survival rate at 18 and 36 months
- Time to initial dose reduction of afatinib
- Proportion of patients with dose modifications of afatinib

# 3.3 Safety Outcome

NA.

#### 4. STUDY DESIGN

# 4.1 General Description

This study was designed as a non-interventional, multi-centre study from existing data of patients who were treated with afatinib in the first-line setting in each study site after the launch of Giotrif® on 7 May 2014 on a regular basis. In first round of data extraction, the data will be extracted retrospectively once patients are enrolled into this study. A second round of data extraction for additional follow-up will be performed one year after completion of first round data extraction.

#### 4.2 Schedule of Events

The schedule of events can be found in Section 6 of the protocol.

Document: \jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018



| Milestone | Planned Date |
|---|---|
| Start of data extraction | Q1 2021 |
| End of data extraction | Q3 2022 |
| Registration in University | Register number not yet assigned as the study is not yet |
| hospital Medical | registered. The study will be registered shortly before |
| Information Network | the start of data extraction. |
| (UMIN) | |
| Final report of study results | Q4 2022 |

# 4.3 Changes to Analysis from Protocol

The following changes were made in this SAP.

- Additional subgroups will be explored in the subgroup analysis. Refer to Section 8.3 for the subgroups to be analyzed.
- All the analyses other than patient disposition and subgroup analysis by initial dose of afatinib will be repeated for patients who initiated afatinib 40mg as first-line setting.

## 5. PLANNED ANALYSES

# 5.1 Interim Analysis

The following data will be analyzed in the interim analysis.

 Document:
 \jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text

 Author:
 Version Number:
 1.0

 Version Date:
 07 DEC 2022

Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018



#### Statistical Analysis Plan

- Patient disposition (participating facilities, reasons for exclusion, etc.)
- Demographics
- Disease characteristics (stage / pathology, type of EGFR gene mutation, etc.)
- Treatment for NSCLC (first-line treatment regimen, second-line treatment regimen, treatment period, reason for treatment discontinuation)
- Outcomes described in Sections 3.1 and 3.2 other than OS and survival rate

# 5.2 Final Analysis

The following data will be analyzed in the final analysis.

• OS and survival rate described in Section 3.2.

## 6. ANALYSIS SETS

## 6.1 All Subjects Enrolled [ENR] Set

The all subjects enrolled (ENR) set will contain all subjects who provide informed consent for this study. This will be used for the analysis of patient disposition.

# 6.2 Analysis Set

The analysis set will contain all enrolled subjects who fulfil all the inclusion criteria and do not present with any of the exclusion criteria. This will be used for all analyses other than patient disposition.

Document: \\jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text

Author: Version Number:


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018 All rights reserved. The contents of this document are confidential and proprietary to its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

1.0



Statistical Analysis Plan

All the analyses other than patient disposition and subgroup analysis by initial dose of afatinib will be repeated for patients who initiated afatinib 40mg as first-line setting.

### 7. GENERAL CONSIDERATIONS

## 7.1 Censoring rule

Censoring rule for time-to-event outcomes is described below.

- ToT1: If patients did not discontinue first-line treatment with afatinib and did not die at the data extraction, they will be censored on the date they are last verified to have been on first-line treatment with afatinib.
- ToT: If patients did not discontinue second-line treatment and did not die at the data extraction, they will be censored on the date they are last verified to have been on second-line treatment. If patients were on first-line treatment and did not move to second-line treatment at the data extraction, ToT is same as ToT1 for these patients.
- ToT2: If patients did not discontinue second-line treatment and did not die at the data extraction, they will be censored on the date they are last verified to have been on second-line treatment.
- OS: If patients did not die at the data extraction, they will be censored on the date they are last verified to be alive.
- Time to initial dose reduction of afatinib: If patients did not reduce initial dose of afatinib at the data extraction, they will be censored on the date they are last verified to have been on the initial dose of afatinib or increased dose of afatinib.

 Document:
 \jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text

 Author:
 Version Number:
 1.0

 Version Date:
 07 DEC 2022

Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

#### 7.2 Software Version

All analyses will be performed using SAS® Software version 9.4 (32bit) or higher.

#### 8. STATISTICAL CONSIDERATIONS

#### 8.1 Statistical Tests and Confidence Intervals

A two-sided 95% confidence interval (CI) will be considered as a default (alpha= 5%). Statistical tests will not be performed.

# 8.2 Missing data

Missing data will not be imputed for the analysis of demographic and disease characteristics described in Section 5.1. Missing data imputation for time-to-event outcomes such as TOT and OS is described in Section 7.1.

# 8.3 Examination of Subgroups

The subgroup categories described below may be modified, depending upon the numbers of patients observed in each subgroup. Some subgroup analyses might not be performed for categories with few patients.

#### Subgroups:

- Patient and disease characteristics
  - Age at the initiation of first-line treatment (>=75 years, <75 years) [Outcomes analysed: TOT1, TOT]</li>
  - EGFR mutation status at the first diagnosis of NSCLC

Document: \iptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

- common, uncommon [Outcomes analysed: TOT1, TOT, OS, Time to initial dose reduction of afatinib]
- each mutation type (Del19, G719X, S768I, L858R, L861Q, Exon 20 insertion, Other) [Outcomes analysed: TOT1, TOT, OS, Time to initial dose reduction of afatinib]
- T790M, Exon 20 insertion, Uncommon mutation other than T790M and Exon 20 insertion [Outcomes analysed: TOT1, TOT, OS, Time to initial dose reduction of afatinib]
- $\circ$  ECOG PS at the initiation of first-line treatment (0/1, >=2) [Outcomes analysed: TOT1, TOT, OS, Time to initial dose reduction of afatinib]
- O Brain metastases at the initiation of first-line treatment (Yes, No) [Outcomes analysed: TOT1, TOT, OS, Time to initial dose reduction of afatinib]
- EGFR mutation status at the initiation of second-line treatment
  - o common, uncommon [Outcomes analysed: TOT, TOT2]
  - o each mutation type (Del19, G719X, S768I, L858R, L861Q, Ins 20, Other) [Outcomes analysed: TOT, TOT2]
  - o T790M, Exon 20 insertion, Uncommon mutation other than T790M and Exon 20 insertion [Outcomes analysed: TOT, TOT2]
- Type of treatment class for subsequent treatment in second-line setting [Outcomes analysed: TOT, TOT2]
- Initial dose of afatinib (Patients starting afatinib 40 mg will be analysed) [Outcomes analysed: TOT1, TOT2, TOT, OS]

# 9. OUTPUT PRESENTATIONS

Continuous variables

Continuous variables will be presented as mean, median, minimum, maximum, Q1, Q3, and standard deviation.

Categorical variables

Categorical variables will be presented as absolute and relative frequency.

Dates & Times

Document: \\jptok-sfs02\\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text


Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018

Copyright © 2018

All rights reserved. The contents of this document are confidential and proprietary to ... and

its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Depending on data available, dates and times will take the form yyyy/mm/dd

Listings

All listings will be ordered by the following (unless otherwise indicated in the template): subject ID, record ID

#### **DISPOSITION AND WITHDRAWALS** 10.

Patients disposition in Section 5.1 will be presented for All Subjects Enrolled Set.

### DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

The descriptive statistics are planned for the following demographic and disease characteristics.

- Age (years) calculated relative to the day of the first dose of Afatinib as first-line treatment
- Sex
- ECOG PS at the initiation of first-line treatment
- Race
- Height (cm) at the initiation of first-line treatment
- Weight (kg) at the initiation of first-line treatment
- Body mass index (BMI) (kg/m<sup>2</sup>) at the initiation of first-line treatment
- Smoking status at the initiation of first-line treatment
- Smoking history (years) at the initiation of first-line treatment
- Smoking history (number/day) at the initiation of first-line treatment
- Period from the day of first diagnosis of NSCLC to the day of the first dose of Afatinib as first-line treatment (month)

\\jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text Document: Author: Version Number: 1.0 Version Date: 07 DEC 2022 Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI WI BIOS0015 Effective Date: 15Jun2018

- Tumor histology at the initiation of first-line treatment
- Type of EGFR mutation at the first diagnosis of NSCLC
- Stage of disease at the initiation of first-line treatment
- Presence of any metastases at the initiation of first-line treatment
- Sites of any metastases at the initiation of first-line treatment
- Treatment with EGFR-TKI before first-line treatment with Afatinib
- Type of EGFR-TKI before first-line treatment with Afatinib
- Period from the end date of EGFR-TKI treatment to the day of the first dose of Afatinib as first-line treatment (year)

#### 11.1 Derivations

• BMI  $(kg/m^2)$  = weight (kg)/ height  $(m)^2$ 

# 12. STUDY MEDICATION EXPOSURE

The descriptive statistics are planned for the data on the treatment for NSCLC.

#### 12.1 Derivations

Duration of exposure to a fatinib as first-line treatment (days) = Cumulative of (Stop date – Start date +1, where daily dose  $\neq 0$ )

Total dose of a fatinib therapy (mg) = Cumulative of daily dose  $\times$  (Stop date – Start date +1).

Duration of off-treatment period for a fatinib therapy (days) = Cumulative of (Stop date – Start date +1, where daily dose = 0).

 Document:
 \jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text

 Author:
 Version Number:
 1.0

 Version Date:
 07 DEC 2022

Template No.: RWI\_TP\_BIOS0013 Revision 1 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Jun2018



# 13. IF AFATINIB THERAPY IS ONGOING AND 'STOP DATE' IS BLANK, THEN 'LAST CONFIRMATION DATE' IS USED AS 'STOP DATE'. OUTCOMES

#### 13.1 **Primary outcome**

The derivation of primary outcome is described in Section 7.1.

Primary outcome will be analysed using Kaplan-Meier method, and the median along with twosided 95% confidence interval (CI) will be displayed (using the Greenwood's formula for estimation of standard errors).

#### 13.2 **Secondary outcomes**

The derivation of time-to event outcomes (TOT, TOT2, OS and time to initial dose reduction of afatinib) is described in Section 7.1.

These time-to-event outcomes will be analysed using Kaplan-Meier method, and the median along with two-sided 95% CI will be displayed (using the Greenwood's formula for estimation of standard errors). For OS, survival rate at 18 and 36 months and its two-sided 95% CI will also be displayed.

## **SAFETY OUTCOMES**

NA

#### REFERENCES 15.

NA

\\jptok-sfs02\data1\PROJ\Boehringer\NZA72277\_Biostatistics\Documentation\SAP\SAP\_text Document:

Author: Version Number: 1.0 Version Date: 07 DEC 2022

Reference: RWI WI BIOS0015

Template No.: RWI TP BIOS0013 Revision 1

Effective Date: 15Jun2018



Study Title: JAPANESE REAL-WORLD DATA FOR TREATMENT OF AFATINIB (GIOTRIF®) IN FIRST-LINE SETTING AND SUBSEQUENT THERAPIES FOR PATIENTS WITH ADVANCED EGFR MUTATION-POSITIVE LUNG ADENOCARCINOMA

**Study Number: 1200-0322** 

**Protocol Version: 1.0** 

I herewith certify that I agree to the content of the study SEAP and to all documents referenced in the study SEAP.

| Position: NIS | | C DocuSigned by | |
|---|---|---|---|
| 1 osition. 1415 | Name/Date: 2022年12月7日 | | この文書を確認した<br>December 7, 2022 5:57:54 AM CET |
| | | Signature: | |
| Position: Global<br>TM Epi | Name/Date: | Signature: | |
| Position: NIS data | Name/Date: | <u></u> | |
| | | Signature: | |
| Position: RWE CoE | Name/Date: | Signature: | |
| | <del>-</del> | | |
| | x-sfs02\data1\PROJ\Boehringer\NZ | A72277_Biostatistics\Documentation\SAF | |
| Template No.: RWI_TF | P_BIOS0013 Revision 1 | Reference: | RWI_WI_BIOS0015 |
| Effective Date: 15Jun2 | 018 | | |
| Copyright © 2018 All | I rights reserved. The contents of this | s document are confidential and proprietary | to . and |

its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

# 完了証明書 エンベロープID: E24601A0895942C8B64FC95C2E6B282F ステータス: 完了 件名: DocuSignで送信: SAP\_NZA72277\_V1.0\_20220107(fix).pdf Project Code (Enter 0 for non-billable projects): 0 ID (Login ID): **Business Unit:** None of the above ソースエンベロープ: 文書ページ数: 18 署名: 2 エンベロープ差出人: 証明書ページ数:5 イニシャル: 0 自動ナビゲーション: 有効 エンベロープIDスタンプ: 無効 タイムゾーン: (UTC+09:00) 大阪、札幌、東京 IPアドレス: レコードの追跡 ステータス: オリジナル 保持者: 場所: DocuSign 2022/12/06 20:28:40 署名者イベント タイムスタンプ 署名 送信: 2022/12/06 20:38:30 表示: 2022/12/06 20:38:44 L-Q STL 署名: 2022/12/06 20:39:27 - Default Part 11 署名の選択: 事前選択のスタイル セキュリティレベル: メール, アカウント認証(必須) 署名ID: 使用IPアドレス: 162.44.230.200 DocuSignパスワードによる署名認証 署名の理由付き(各タブ上): この文書を承認する 電子記録および電子署名の開示条件: DocuSignで設定されていません NBI 水島 送信: 2022/12/06 20:39:30 表示: 2022/12/06 20:55:56 セキュリティレベル: メール, アカウント認証(必須) 署名: 2022/12/06 20:58:03 署名の選択: 事前選択のスタイル 署名ID:

使用IPアドレス: 165.225.97.71

DocuSignパスワードによる署名認証

署名の理由付き(各タブ上): この文書を確認した

電子記録および電子署名の開示条件:

同意: 2022/12/06 20:55:56

| 同席署名者イベント | 署名 | タイムスタンプ |
|------------------|------------|---------------------|
| 編集者配信イベント | ステータス | タイムスタンプ |
| 代理人配信イベント | ステータス | タイムスタンプ |
| 仲介者配信イベント | ステータス | タイムスタンプ |
| 証明書付き配信イベント | ステータス | タイムスタンプ |
| カーボンコピーイベント | ステータス | タイムスタンプ |
| 立会人イベント | 署名 | タイムスタンプ |
| 公証人イベント | 署名 | タイムスタンプ |
| エンベロープ概要イベント | ステータス | タイムスタンプ |
| エンベロープの送信 | ハッシュ/暗号化済み | 2022/12/06 20:38:30 |
| 証明書付き配信 | セキュリティ確認済み | 2022/12/06 20:55:56 |
| 署名の完了 | セキュリティ確認済み | 2022/12/06 20:58:03 |
| 完了 | セキュリティ確認済み | 2022/12/06 20:58:03 |
| 支払いイベント | ステータス | タイムスタンプ |
| 電子記録および電子署名の開示条件 | | |

| CONSENT TO ELECTR | . / | <br>17373747171171171317 |
|-------------------|-----|--------------------------|

From time to time, ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

# **Documents will be sent to you electronically**

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

# Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

# **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

# How to contact

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact:

1. To advise of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to a like the sent to a different e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

| 2. To request paper copies from | | |
|---|---|---|
| To request paper copies of Documents y | ou have received previously through y | our DocuSign |
| user account send an e-mail to | | |

user account, send an e-mail to

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii)
U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

# 3. To withdraw your consent with

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

# Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

## Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify as as described above, you consent to the delivery and execution of Documents electronically.